CLINICAL TRIAL: NCT05157750
Title: Direct Comparison of Endoscopic and Histologic Remission and Barrier Healing for Predicting Long Term Disease Behaviour in Clinically Remittent IBD Patients: the Prospective ERIca Study
Brief Title: Endoscopic Remission, Histologic Remission and Barrier Healing for Predicting Disease Behaviour in IBD
Acronym: ERIca
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Timo Rath, Professor for Endoscopy, Consultant in Gastroenterology, University of Erlangen-Nürnberg Medical School
Other Study IDs: ERIca Study
Record Dates: First submitted 2021-10-19; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IBD patients with endoscopic remission: No intervention will be administered. All patients with endoscopic remission will be monitored for the future development of major clinical events. Diagnostic performances of endoscopic remission for predicting major clinical events will be calculated.
  Interventions: Other: Recording of major clinical events
- IBD patients with histologic remission: No intervention will be administered. All patients with histologic remission will be monitored for the future development of major clinical events. Diagnostic performances of histologic remission for predicting major clinical events will be calculated.
  Interventions: Other: Recording of major clinical events
- IBD patients with barrier healing: No intervention will be administered. All patients with barrier healing will be monitored for the future development of major clinical events. Diagnostic performances of barrier healing for predicting major clinical events will be calculated.
  Interventions: Other: Recording of major clinical events

INTERVENTIONS:
Other: Recording of major clinical events — During follow-up, major clinical events, defined as (i) disease flare; (ii) IBD-related hospitalization, (iii) IBD-related surgery, (iv) necessity for initiation of systemic steroids, immunosuppressants or biologics; (v) necessity for escalation of an existing biological therapy, will be recorded.

SUMMARY:
Within this study, the investigators aim to directly compare the value of endoscopic remission, histologic remission and barrier healing for predicting long-term disease behavior in a large cohort of clinically remittent IBD patients.

DETAILED DESCRIPTION:
Mucosal healing is a key therapeutic goal in the management of patients with inflammatory bowel diseases (IBD) that is associated with favorable long-term disease outcome. In addition, histologic remission is an emerging endpoint and first data suggest that functional assessment of the integrity of the intestinal barrier, i.e. barrier healing, by confocal laser endomicroscopy (CLE) correlates to clinical disease behavior and outcome.

Within this study, the investigators will prospectively include IBD patients in clinical remission and assess endoscopic remission, histologic remission and barrier healing during baseline ileocolonoscopy. Participants will then be closely followed up in the IBD outpatient department of the University Hospital Erlangen every 4 to 8 weeks for participants under biological therapy and every 8 weeks for participants under conventional therapy. At each visit, clinical disease activity using the Mayo Clinical Score (MCS) and the Crohn's disease activity Index (CDAI), respectively, routine laboratory parameters and current and past medications will be recorded. Further, at each visit, major clinical events (MCE), defined as (i) disease flare; (ii) IBD-related hospitalization, (iii) IBD-related surgery, (iv) necessity for initiation of systemic steroids, immunosuppressants or biologics; (v) necessity for escalation of an existing biological therapy, will be recorded. The primary endpoint of this study is to comparatively assess the predictive values of barrier healing, endoscopic remission and histologic remission for predicting occurrence of MCE in IBD patients in clinical remission

ELIGIBILITY:
Inclusion Criteria:

* patients with an established IBD diagnosis for at least 12 months duration
* IBD patients in clinical remission

Exclusion Criteria:

* patients with poor bowel preparation
* patients with total colectomy,
* patients with concomitant beta blocker therapy,
* patients with known allergy to fluorescein
* patients with a planned change in IBD-related pharmacotherapy

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with an established IBD diagnosis for at least 12 months duration presenting in clinical remission presenting at the Department of Gastroenterology of the University Hospital Erlangen will be prospectively included.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-01-16 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of endoscopic remission in ulcerative colitis | 2 years
  Endoscopic remission will be assessed using the Mayo Endoscopy Score in ulcerative colitis
Predictive value of endoscopic remission in Crohn's disease | 2 years
  Endoscopic remission will be assessed using the simplified endoscopic index of severity (SES-CD) in Crohn's disease
Predictive value of histologic remission in ulcerative colitis | 2 years
  Histologic remission will be assessed using the Robarts Histology Index and the Nancy Histology Index in ulcerative colitis
Predictive value of histologic remission in Crohn's disease | 2 years
  Histologic remission will be assessed using a modified Riley Score in Crohn's disease
Predictive value of barrier healing | 2 years
  Barrier healing will be assessed using the well-established Watson-Score as a semiquantitative grading system of the intestinal barrier function

CONTACTS AND LOCATIONS:
Overall Officials: Timo Rath, MD, Principal Investigator — University Hospital Erlangen, Department of Medicine 1
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rath T, Atreya R, Bodenschatz J, Uter W, Geppert CI, Vitali F, Zundler S, Waldner MJ, Hartmann A, Neurath MF. Healing of the epithelial barrier in the ileum is superior to endoscopic and histologic remission for predicting major adverse outcomes in ulcerative colitis. Front Med (Lausanne). 2023 Oct 10;10:1221449. doi: 10.3389/fmed.2023.1221449. eCollection 2023. PMID 37881628
- [Derived] Rath T, Atreya R, Bodenschatz J, Uter W, Geppert CE, Vitali F, Fischer S, Waldner MJ, Colombel JF, Hartmann A, Neurath MF. Intestinal Barrier Healing Is Superior to Endoscopic and Histologic Remission for Predicting Major Adverse Outcomes in Inflammatory Bowel Disease: The Prospective ERIca Trial. Gastroenterology. 2023 Feb;164(2):241-255. doi: 10.1053/j.gastro.2022.10.014. Epub 2022 Oct 21. PMID 36279923